CLINICAL TRIAL: NCT03045185
Title: A Prospective Clinical Study of Regenerative Endodontic Treatment of Traumatised Non-vital Immature Teeth Using Bi-antibiotic Paste
Brief Title: Regenerative Endodontic Treatment of Traumatised Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Hani Nazzal, Dr, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC 12/YH0488
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Tooth Injuries; Endodontically Treated Teeth
Keywords: Non Vital teeth; Traumatised teeth; Immature teeth; Regenerative Endodontics
MeSH Terms: conditions — Tooth Injuries; Tooth, Nonvital | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Prospective interventional uncontrolled trial
Masking Description: Single group so no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): RET using Ciprofloxacin 100mg, and Metronidazole 100mg.
  Interventions: Procedure: RET using Ciprofloxacin 100mg, and Metronidazole 100mg.

INTERVENTIONS:
Procedure: RET using Ciprofloxacin 100mg, and Metronidazole 100mg. — First Treatment Visit: Tooth isolation, access, pulp extirpation and root canal irrigation with 0.5% sodium hypochlorite. Canal negotiation, canal drying using paper points. Delivery of the Bi antibiotic paste (mixture of Bi antibiotic paste (Ciprofloxacin 100mg and Metronidazole 100mg with sterile water). Sealing tooth access with glass ionomer cement.
  Second Treatment Visit: Tooth analgesia using plain local analgesics, isolatation and re-access as described above. Irrigation of root canal system using normal saline followed by paper point dying. Initiation of bleeding through insertion of a sterile 23-gauge needle with a length of 2 mm beyond the working length into the periapical tissues. Access sealed using Portland cement, followed by glass ionomer and then composite resin.

SUMMARY:
Aim: The aim of this prospective study was to evaluate the treatment outcomes of regenerative endodontic technique (RET) for the management of traumatised non-vital immature teeth in children. Methodology: This study aims to recruit 25-30 healthy children with traumatised non-vital immature upper incisors to be treated with bi-antibiotic regenerative endodontic technique. Patients will be reviewed clinically at 3m,6m,9m,12m,2y,and 3 years and radiographically at 3m,9m, 2y,and 3 years. One operator will undertake all treatments, clinical reviews and standardised radiographic exposures. Radiographic analysis will be carried out by two calibrated experienced clinicians. Standardised photographs will be taken at 3m,12m,2y,and 3 years and crown colour changes will be assessed using a standardised validated methodology.

DETAILED DESCRIPTION:
Aims of the pilot study:

Primary:

* Study the clinical and radiographic success of Regenerative Endodontic Technique for the regeneration/revascularisation of immature permanent teeth with necrotic root canal systems following a traumatic injury.
* Study the qualitative and quantitative increase in root dimensions, following RET, by evaluating continued root development and thickening of dentinal walls.

Secondary:

Evaluate effect of treatment on colour change of the treated tooth compared with the healthy contralateral tooth.

Hypothesis:

Through the repopulation of the root canal space with vital tissue, Regenerative Endodontic Technique would promote continued root development and/or thickening of the dentinal walls, thereby improving the long-term prognosis of non vital immature traumatised teeth.

Methodology:

Design of the pilot study:

This will be a prospective interventional study.

Participants:

This study aims to recruit 25-30 patients. This estimation is based on discussion with the statistician and an estimation of the number of children who are referred to the LDI with non-vital immature anterior teeth following trauma, who might be eligible for participation in the study. Ethical approval will be sought through the Integrated Research Application System (IRAS). Patients referred to the Paediatric Dentistry Department at the Leeds Dental Institute (LDI) will be assessed by the clinicians for suitability for inclusion into this study based on the following inclusion and exclusion criteria.

Intervention:

At the RET clinic and once an informed consent is obtained, the treatment will be carried out over two visits each lasting about 45 minutes. During these visits, patients received the following treatment:

First Treatment Visit:

* Preoperative photographs will be taken by the principal investigator using a Fujifilm (Tokyo, Japan), Finepix S3 Pro camera with 105-mm Micro Nikon (Tokyo, Japan) f2.8 lens and sigma ring flash, EM-140DG.
* The tooth will be isolated using dry dam (Directa, Upplands Visby, Sweden).
* The tooth will be accessed and the pulp will be extirpated. The root canal system will then be irrigated with copious chemical disinfectant ( 0.5% sodium hypochlorite) for 15 minutes.
* The canal will then be negotiated with minimal or no filing to prevent further weakening of the existing dentinal walls.
* The canal will then be dried using paper points.
* In an ante-room, the two antibiotics, Ciprofloxacin and Metronidazole, will be mixed with sterile water.
* The mixture of the two antibiotics will then be carried into the root canal with special applicators so that the entire root canal is filled with the antibiotics.
* The root canal will then be hermetically sealed with a glass ionomer cement to prevent any coronal leakage or contamination of the root canal with oral microorganisms. The patient will then be discharged and an appointment made for two weeks later.

Second Treatment Visit:

* Local analgesia will be administered and the tooth will be isolated and re-accessed as described above.
* The antibiotic mixture will be flushed out of the root canal by irrigation with normal saline. Following this the root canal will be thoroughly dried with paper points.
* This will then be followed by insertion of a sterile 23-gauge needle with a length of 2 mm beyond the working length and past the confines of the root canal into the periapical tissues to intentionally induce bleeding into the root canal. The bleeding is then allowed to fill the root canal.
* Once the root canal is filled with blood, a cotton pledget will be placed in the pulp chamber and a clot will be allowed to form in the root canal.
* Once the clot has formed the pulp chamber in the coronal part will be thoroughly cleaned to remove any remnants of the blood, which could cause discolouration in the future.
* The access cavity will then be hermetically sealed with three layers of material to prevent coronal leakage and contamination; Portland cement, followed by glass ionomer and then composite resin.
* Patients will then be reviewed after 3, 6 and 9 months.

Review visits and outcomes The patients will be reviewed after 3, 6, 9 and , 12 months, 2 years and 3 years.

The following outcomes will be assessed:

Clinical:

The following will be assessed:

* Presence of normal physiologic tooth mobility.
* Tenderness to percussion.
* Free from pain or discomfort.
* No evidence of labial swelling signifying continued presence of infection.

Radiographic:

Standardised periapical radiographs will be taken before start of treatment, during the treatment and then again at 3 months,and after 9 months, 2 years and 3 years.

Trained independent examiners:

Two trained and independent examiners will evaluate the radiographs. All radiographs will be randomly shown to the examiners who will be independently asked to score the test parameters.

Image analysis:

Continuous root development, changes in dentinal root thickness and apical foramen width will be quantified.

Pulp Sensibility Tests:

At each recall pulp sensibility responses will be evaluated using thermal test (Ethyl Chloride) and Electric Pulp test (EPT).

Photographs:

Standardised intra-oral photographs will be taken before start of the treatment, 9-month, 2 years, and 3 years follow-up visits. Favourable post treatment crown colour in comparison to the pre operative photographs and to that of the contralateral tooth will be assessed using the MathWorks software as described in the study by Day et al. in 2011.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6-16 years of age
* Patients who are fit and healthy or with an ASA1 or ASA2 medical conditions
* Patients with cooperation level that would allow treatment under local analgesia
* Patients with a traumatised permanent incisors, canines or premolars having at least one of the following:

  * Necrotic or partially necrotic root canal systems.
  * Periapical periodontitis/abscess.
  * Sinus tract.
* Patients with permanent incisors, canines or premolars that have incomplete root formation with open apices.

Exclusion Criteria:

* Patient older than 16 year of age
* Patients allergic to Ciprofloxacin, Metronidazole.
* Patients with medical conditions and/or receiving medications that would affect patients' body's ability to heal such as diabetic patients or ability of the patients' blood to clot such as patients with Von Willebrand's disease.
* Patients with risk of developing infective endocarditis or immune compromised patients.
* Patients with non traumatised non-vital permanent incisors, canines or premolars where root development already deemed to be completed.
* No concurrent signs of other pathological root resorption, such as replacement root resorption, which could otherwise affect the prognosis of the tooth.
* Uncooperative patients.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change in root length | Month 3, Month 9, Year 2, and year 3.
  Root length from cement enamel junction to radiographic apex measured over time
Change in root dentinal wall width | Month 3, Month 9, Year 2, and year 3.
  Root dentinal width measured radiographically at 2/3 root length over time
Change in apical foramen width | Month 3, Month 9, Year 2, and year 3.
  Apical foramen width measured radiographically over time
Change in periodontal healing | Month 3, Month 6, Month 9, Year 2, and year 3.
  Absence of signs and symptoms of infection over time

SECONDARY OUTCOMES:
Change in crown Colour | Month 3,Month 12, year 2, and year 3.
  Crown colour change measured using CIELAB scores

CONTACTS AND LOCATIONS:
Overall Officials: Hani Nazzal, BDS, PhD, Principal Investigator — University of Leeds, School of Dentistry, Paediatric Dentistry Department

IPD SHARING:
Plan to Share IPD: No
Not planning on IPD